CLINICAL TRIAL: NCT01715168
Title: A Phase 1, Single-blind, Randomized, Two-way, Crossover Bioequivalence Study of Intravenously Administered ATI 0918 in Patients With Ovarian Cancer That Has Progressed or Recurred After Platinum-based Chemotherapy
Brief Title: A Crossover Bioequivalence Study of Intravenously Administered ATI0918 and DOXIL/CAELYX in Patients With Ovarian Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Azaya Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: ATI0918-101
Record Dates: First submitted 2012-10-19; First posted 2012-10-26 (Estimated); Last update posted 2015-01-15 (Estimated); Status verified 2015-01

CONDITIONS: Ovarian Cancer; Malignant Female Reproductive System Neoplasm; Cancer; Ovarian Tumor; Ovarian Epithelial Cancer Recurrent
Keywords: Doxil generic; Caelyx generic; generic treatment; ovarian cancer; ovary; progressed; recurred cancer; platinum based therapy
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms | interventions — liposomal doxorubicin; Doxorubicin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DOXIL/CAELYX or Doxorubicin Hydrochloride (Lipspome) (Active Comparator): Current Standard of care and/or reference product in Europe (Caelyx) and US (Doxorubicin Hydrochloride (Liposome) and Doxil)
  Interventions: Drug: DOXIL/CAELYX
- ATI-0918 (Experimental): Investigational drug arm which will be compared to Doxil/Caelyx and Hydrochloride Doxorubicin (Liposome) arms for bioequivalence analysis
  Interventions: Drug: ATI-0918

INTERVENTIONS:
Drug: DOXIL/CAELYX
  Other Names: Doxorubicin Hydrochloride; Doxil; Caelyx; Liposomal doxorubicin hydrochloride
  Arms: DOXIL/CAELYX or Doxorubicin Hydrochloride (Lipspome)
Drug: ATI-0918
  Other Names: doxorubicin hydrochloride; liposomal doxorubicin hydrochloride
  Arms: ATI-0918

SUMMARY:
The purpose of this study is to find the answers to the following research question(s):

1. Is the study drug equivalent to the approved drug, Doxil/Caelyx, and does it act the same way in the body as the approved drug?

ATI-0918 is believed to be a generic of Doxil/Caelyx and this is what the study is trying to prove. All people who participate in this study will receive the research study medication (ATI-0918) and Doxil/Caelyx in addition to best supportive care (treatment for symptoms).

The study drug being tested in this study works the same as the FDA (government) approved drug doxorubicin HCl. ATI-0918 is a generic (the same) formulation of doxorubicin HCl being delivered (given to the patient).

ELIGIBILITY:
Inclusion Criteria:

1. Have histologically confirmed ovarian cancer that is potentially sensitive to DOXIL/CAELYX
2. Have disease progression or recurrence after a maximum of 2 prior chemotherapies, one of which was platinum based.
3. Be DOXIL/CAELYX treatment naïve
4. Have a normal left ventricular ejection fraction (LVEF) based on institutional ranges.
5. Have an Eastern Cooperative Oncology Group (ECOG) performance status of </= 2
6. Have an estimated life expectancy of ≥ 3 months
7. Be >/= 18 and </= 70 years of age
8. Sign a written Institutional Review Board (IRB)-approved informed consent form
9. Have a negative pregnancy test, if patient is of child-bearing potential
10. Have acceptable liver function:

    * Bilirubin </= upper limit of normal (ULN)
    * AST (SGOT), ALT (SGPT) and Alkaline phosphatase </= 1.5 times upper limit of normal
11. Have acceptable renal function:

    * Serum creatinine within normal limits, OR calculated creatinine clearance >/= 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
12. Have acceptable hematologic status:

    * Neutrophils >/= 1500 cells/mm3
    * Platelet count >/= 100,000 (plt/mm3)
    * Hemoglobin >/= 9 g/dL
13. Have acceptable coagulation status:

    * Prothrombin time (PT) or International Normalized Ratio (INR) within 1.5 × ULN
    * Partial thromboplastin time (PTT) within 1.5 × ULN
14. Agree to use effective contraceptive methods during the study (nonsterile patients of childbearing potential)

Exclusion Criteria:

1. Have New York Heart Association (NYHA) Class III or IV cardiac disease, myocardial infarction within the past 6 months prior to Day 1, unstable arrhythmia, or evidence of ischemia on electrocardiogram (ECG) or during Cardiac Stress Testing within 14 days prior to Day 1
2. Have received > 250 mg/m2 of doxorubicin or equivalent as other anthracyclines or similar compounds
3. Have received prior treatment with DOXIL/CAELYX
4. Have received radiotherapy to the mediastinal area or concomitant therapy with other potentially cardiotoxic agents
5. Have seizure disorders requiring anticonvulsant therapy
6. Have known brain metastases (unless previously treated and well controlled for a period of >/= 3 months)
7. Have severe chronic obstructive pulmonary disease with hypoxemia
8. Have had major surgery, other than diagnostic surgery, within 4 weeks prior to Day 1
9. Have an active, uncontrolled bacterial, viral, fungal, or other opportunistic infections requiring systemic therapy
10. Are pregnant or nursing. NOTE: Nonsterile women of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; or abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
11. Have received treatment with radiation therapy, surgery, chemotherapy, or investigational therapy within one month prior to study entry (6 weeks for nitrosoureas or Mitomycin C).
12. Have received radiation therapy to >25% of her total bone marrow during her lifetime
13. Are unwilling or unable to comply with procedures required in this protocol
14. Have known infection with human immunodeficiency virus (HIV), hepatitis B, or hepatitis C
15. Have a serious nonmalignant disease (e.g., hydronephrosis, liver failure, significantly impaired hepatic function, or other conditions) that could compromise protocol objectives in the opinion of the investigator and/or the sponsor
16. Are currently receiving any other investigational agent
17. Have exhibited allergic reactions to doxorubicin or a similar structural compound

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-10; Primary Completion 2015-10 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of AUC in a single dose of ATI0918 vs single dose of Doxil/Caelyx | pre, 30 min + pre, 0, .50, 1, 2, 4, 6, 24, 48, 72, 120, 168, 216 hour post infusion for 2 Cycles (Cycle is defined as 28 days)
  The primary objective of this study is to determine the pharmacokinetic equivalence of ATI-0918 and DOXIL/CAELYX as a single dose in patients with ovarian cancer. The outcome measure will be determined by analyzing PK data from drawn from each patient at pre-specified time points and calculating Area under the curve (AUC) and Peak Plasma Concentration (Cmax)to determine % variability between ATI0918 and Doxil/Caelyx within each patient.
Comparison of Cmax in a single dose of ATI0918 vs single dose of Doxil/Caelyx | pre, 30 min + pre, 0, .50, 1, 2, 4, 6, 24, 48, 72, 120, 168, 216 hour post infusion for 2 Cycles (Cycle is defined as 28 days)
  The primary objective of this study is to determine the pharmacokinetic equivalence of ATI-0918 and DOXIL/CAELYX as a single dose in patients with ovarian cancer. The outcome measure will be determined by analyzing PK data from drawn from each patient at pre-specified time points and calculating Area under the curve (AUC) and Peak Plasma Concentration (Cmax)to determine % variability between ATI0918 and Doxil/Caelyx within each patient.

CONTACTS AND LOCATIONS:
Locations (2):
- Yakima Valley Memorial Hospital - North Star Lodge, Yakima, Washington, United States
- Centre Hospitalier de L'Universite de Montreal (CHUM), Montreal, Quebec, Canada